CLINICAL TRIAL: NCT02135562
Title: A Pilot Study of a Protein-Sparing Modified Fast for Weight Loss in Obese Endometrial Cancer Survivors
Brief Title: Protein-Sparing Modified Fast Intervention for Weight Loss in Obese Endometrial Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1814; NCI-2014-00832 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE1814; CASE 1814 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Endometrial Cancer; Obesity
Keywords: endometrial cancer; survivor; obesity; diet; high protein; protein-sparing modified fast intervention; PSMF
MeSH Terms: conditions — Endometrial Neoplasms; Obesity | interventions — Diet Therapy; Nutrition Assessment; Methods; Body Weight Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (PSMF) (Experimental): Participants will take part in a Protein-Sparing Modified Fast (PSMF) Intervention for weight loss. Participants will undergo a dietary intervention high in protein for 6 weeks or until they have loss 15% of their body weight. This intervention will be followed by weight maintenance in which participants reintroduce non-starchy vegetables to their diet. At this time participants will also receive informational material and dietary education which teaches participants how to read nutrition labels and calculate carbohydrate loads in foods. Participants are given the Obesity and Weight-Loss Quality of Life Questionnaire to survey the impact of the intervention
  Interventions: Dietary Supplement: Dietary Intervention; Other: Informational Material; Other: Dietary Education; Dietary Supplement: Weight Maintenance; Other: Average score of Obesity and Weight-Loss Quality of Life Questionnaire

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — Follow the Protein-Sparing Modified Fast (PSMF) intervention. This diet has participants consume enough lean beef, pork, poultry, and seafood to provide 1.2 grams of protein per kilogram of their obesity adjusted ideal body weight.
  Other Names: Dietary Modification; intervention, dietary
Other: Informational Material — Receive carbohydrate reintroduction handout
Other: Dietary Education — Receive education on nutrition label reading for carbohydrates
  Other Names: intervention, educational
Dietary Supplement: Weight Maintenance — weight maintenance diet consists of gradual addition of previously eliminated carbohydrate containing food groups to the high protein PSMF diet. During weight maintenance, consumption of non-starchy vegetables is unlimited
Other: Average score of Obesity and Weight-Loss Quality of Life Questionnaire — Participants will take a tailored quality of life questionnaire. These scores will be averaged and a group mean reported. Higher scores indicate greater quality of life.

SUMMARY:
This pilot clinical trial studies protein-sparing modified fast (PSMF) intervention for weight loss in obese endometrial cancer survivors. The PSMF is a diet that is very low in carbohydrates and calories, designed to induce fast, safe weight loss. The diet consists of only lean meats (beef, pork, poultry, and seafood) in amounts adequate to meet protein requirements based on the individual's body weight. The PSMF may help endometrial cancer survivors achieve significant weight loss, reduce the risk of chronic disease, and improve quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Investigate whether the PSMF leads to significant weight loss in obese endometrial cancer survivors (ECS).

II. To assess whether the approach is feasible, whether participants will remain in the study for the duration of the intervention while adhering to the various components of the protocol. To assess feasibility, examine the following variables: drop-out rates; rates of adherence to diet and supplemental protocol; and rates of common side-effects.

III. Assess whether the PSMF improves biomarkers of disease risk in this population. To assess whether this objective has been met, assess the following variables: blood lipids (total cholesterol, low density lipid [LDL] cholesterol, high density lipid [HDL] cholesterol, and triglycerides); glucose; and markers of inflammation (C-reactive protein, interleukin-6, tumor necrosis factor [TNF]-alpha, and leptin).

IV. Assess whether the PSMF leads to improvement in quality of life related to weight loss.

OUTLINE:

PSMF: Participants are instructed by a registered dietitian (RD) to consume enough lean beef, pork, poultry, and seafood to provide 1.2 grams of protein per kilogram of their obesity adjusted ideal body weight. The protein recommendation will be communicated to participants in terms of grams per day. Participants are encouraged to adhere as closely as possible to the protein recommendation. Based on the protein recommendation, participants are advised to consume a given amount (in ounces) of beef, pork, poultry and seafood daily, assuming that each ounce of these products contains seven grams of protein. Participants are provided with a digital kitchen scale to weigh protein-containing foods and are permitted up to 2 servings of non-starchy vegetables per day. Participants remain on the PSMF until they have successfully reduced their initial body weight by 15% or up to 6 months. Participants are also provided with supplements to consume daily.

WEIGHT MAINTENANCE DIET: After successful weight loss of at least 15% of initial body weight, participants are instructed by a RD to consume a weight maintenance diet or they may remain on the PSMF. The weight maintenance diet consists of gradual addition of previously eliminated carbohydrate containing food groups to the PSMF and consumption of non-starchy vegetables is unlimited. Participants receive handouts that list common foods and the number of carbohydrates in each serving and educated on nutrition label reading for carbohydrates, with emphasis on serving size and total number of carbohydrates per serving.

After completion of study, participants are followed up at 2 and 4 weeks and then at 2, 3, 4, 5, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of endometrial cancer, successfully treated through surgery
* Body mass index (BMI) > 30 kg/m^2
* > 8 weeks removed from surgery to treat endometrial cancer

Exclusion Criteria:

* No previous diagnosis of endometrial cancer
* BMI < 30 kg/m^2
* Any history of cardiovascular, kidney, or liver disease
* Using medication to treat diabetes
* History of cardiac arrhythmias
* Inability to comply with follow up regimen
* Inability to read or speak English
* Abstention from meat and other animal products

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-08-08 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Mean Weight loss assessed with the digital scale | Baseline up to 6 months
  Mean weight loss will be presented as mean total weight loss in kilograms from baseline
Mean Weight loss assessed with the digital scale | Baseline up to 12 months
  Mean Weight loss will be presented as mean total weight loss in kilograms from baseline.

SECONDARY OUTCOMES:
Changes in levels of total cholesterol | Baseline up to 6 months
  Average differences in total cholesterol between time points will be assessed using a one-sided anova test with statistical significance defined as having a p-value < 0.05.
Changes in levels of markers of inflammation (C-reactive protein) | Up to 6 months
  Average differences in C-reactive protein between time points will be assessed using a one-sided anova test with statistical significance defined as having a p-value < 0.05.
Changes in levels of glucose | Up to 6 months
  Differences in glucose levels between time points will be assessed using a one-sided anova test with statistical significance defined as having a p-value < 0.05.
Number of drop-out participants | Up to 6 months
  Presented as the difference in the number of participants who completed the study from the number of participants enrolled at baseline. This is reported as one of the markers of feasibility.
Average percentage of positive urinary ketone tests as a marker of dietary adherence | Up to 6 months
  Assessed using the presence of urinary ketones beginning on day four of the intervention. Adherence rates will be presented as the percentage of positive urinary ketone tests for the duration of the intervention.
Number of Participant with reported side effects | Up to 6 months
  Adverse events will be recorded by participants on a daily basis. Number of participants with related adverse events will be reported as one of the measures of feasibility
Changes in quality-of-life as assessed by the Obesity and Weight Loss Quality-of-Life Questionnaire | Baseline up to 6 months
  The difference between mean quality of life scores at the two time points will be assessed using a one-sided anova test with statistical significance set at p < 0.05.
Changes in levels of markers of inflammation (interleukin 6) | Up to 6 months
  Average differences in interleukin 6 between time points will be assessed using a one-sided anova test with statistical significance defined as having a p-value < 0.05.
Changes in levels of markers of inflammation (tumor necrosis factor - alpha) | Up to 6 months
  Average differences in tumor necrosis factor - alpha between time points will be assessed using a one-sided anova test with statistical significance defined as having a p-value < 0.05.
Changes in levels of markers of inflammation (leptin) | Up to 6 months
  Average differences of leptin between time points will be assessed using a one-sided anova test with statistical significance defined as having a p-value < 0.05.
Changes in levels of LDL-cholesterol | Baseline up to 6 months
  Average differences between time points for LDL-cholesterol will be assessed using a one-sided anova test with statistical significance defined as having a p-value < 0.05.
Changes in levels of HDL-cholesterol | Baseline up to 6 months
  Average differences between time points for HDL-cholesterol will be assessed using a one-sided anova test with statistical significance defined as having a p-value < 0.05.
Changes in levels of triglycerides | Baseline up to 6 months
  Average differences between time points for triglycerides will be assessed using a one-sided anova test with statistical significance defined as having a p-value < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Resnick, Principal Investigator — Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Cleveland Medical Center, University Hospitals, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio